# STATISTICAL ANALYSIS PLAN

EXTRACT-PE: A Prospective, Multicenter Trial to Evaluate the Safety and Efficacy of the Indigo® Aspiration System in Acute Pulmonary Embolism

**Protocol CLP-11373** 

May 7, 2019

### Contents

| 1 | Ove | Overview4 | |
|---|---|---|---|
| 2 | Sar | nple Size | 4 |
| | 2.1 | Effectiveness Power | 5 |
| | 2.2 | Safety Power | 5 |
| | 2.3 | Justification of Effectiveness and Safety Thresholds | 6 |
| 3 | Inte | erim Analysis | 7 |
| | 3.1 | Re-estimation of Sample Size | 8 |
| 4 | Analysis Populations | | 11 |
| | 4.1 | Definitions | 11 |
| 5 | Sta | tistical Methods | 13 |
| 6 | Bas | seline Characteristics | 13 |
| 7 | Pat | ient Disposition | 13 |
| 8 | Effe | ectiveness Analysis | 14 |
| | 8.1 | Primary Effectiveness Analysis | 14 |
| | 8.2 | Handling of Multiplicity | 15 |
| 9 | Sub | ogroup Analysis | 15 |
| 10 | Saf | ety Analysis | 16 |
| | 10.1 | Primary Safety Analysis | 16 |
| | 10.2 | Secondary Safety Analysis | 16 |
| | 10.3 | Analysis of Adverse Events | 17 |
| | 10.4 | Handling of Multiplicity | 17 |
| | 10.5 | Analysis of Deaths | 17 |
| 11 | Pod | oling Across Centers | 18 |
| 12 | Los | t to Follow-Up and Missing Data | 18 |
| 13 | Blin | nding | 19 |
| 14 | Cor | nmittees | 19 |
| | 14.1 | Clinical Events Committee (CEC) | 19 |
| | 14.2 | Data Safety Monitoring Board (DSMB) | 19 |
| | 14.3 | Core Lab | 19 |
| 15 | Cha | anges to Planned Analyses | 19 |

| 16 | Referer | nces | . 20 |
|----|----------|-------------------------------------|------|
| 17 | SAS Co | ode | . 24 |
| 1 | 7.1 Pri | mary Efficacy Power Calculation | . 24 |
| | 17.1.1 | Code | . 24 |
| | 17.1.2 | Output | .24 |
| 1 | 7.2 Priı | mary Safety Power Calculation | . 25 |
| | 17.2.1 | Code | . 25 |
| | 17.2.2 | Output | . 25 |
| 1 | 7.3 Saı | mple Size Re-Estimation Calculation | .26 |

### 1 Overview

This is a prospective multi-center, single-arm study designed to evaluate the effectiveness and safety of the INDIGO<sup>™</sup> Aspiration System for aspiration mechanical thrombectomy in patients with acute pulmonary embolism (PE).

Up to 150 adult patients will be enrolled from approximately 25 centers in order to provide 100 evaluable patients after attrition. Each site will be limited to a maximum enrollment of up to 30 patients (~20% of total enrollment). Depending on an interim sample size review, the number of patients enrolled may increase up to 300 patients in order to provide up to 200 evaluable patients (for further details please refer to section 3.1).

This Statistical Analysis Plan (SAP) will provide details to further elaborate statistical methods as outlined in the protocol and will describe analysis conventions. The SAP will be signed off prior to database lock.

### 2 Sample Size

A sample size of up to 150 enrolled patients was selected for this study in order to provide 100 evaluable patients. Assuming a mean change of 0.42 in the RV/LV ratio from baseline to 48 hours and a standard deviation of 0.36 the two-sided 95% normal distribution confidence interval for a sample size of 100 patients is (0.35, 0.49). The estimated mean and standard deviation are based on clinical data from the SEATTLE II study of pulmonary embolism treatment (Piazza 2015).

Assuming a 48 hour major adverse events rate of 15% (15/100), the two-sided 95% normal distribution confidence interval is (8.0%, 22.0%). This estimated rate is based on complications reported for interventional treatment (Piazza 2015, Kucher 2014, Kuo 2015, Stein 2012, Neely 2015, Aklog 2002, Greenlish, 2011).

To account for up to 33% attrition, the enrollment was increased to 150 patients. The effectiveness and safety sample size calculations support 150 enrolled patients (Table 1 and Table 2).

### 2.1 Effectiveness Power

The effectiveness hypothesis tested is that the mean change in RV/LV ratio from baseline to 48 hours, RV/LV<sub>change</sub>, does not equal 0.2:

 $H_0$ : RV/LV<sub>change</sub> = 0.2

vs  $H_a$ : RV/LV<sub>change</sub>  $\neq$  0.2,

under an observed mean of 0.42 and standard deviation of 0.36 at alpha = 0.05.

The power for a one-group, two-sided test for a single mean difference was calculated for the test using SAS v 9.4 (SAS Institute, Cary, NC). The SAS code and output are provided in Section 17.

Table 1. Effectiveness Sample Size Parameters

| Alpha | 0.05 |
|------------------------------|-----------------------------|
| Sides | 2 |
| Estimated mean | 0.42 |
| Estimated standard deviation | 0.36 |
| Null mean $(\mu_0)$ | 0.2 |
| N | 100 |
| Power | >.999 |
| Attrition | 33% |
| Total N | 100 x 1/(1 - 0.33) =<br>150 |

# 2.2 Safety Power

The safety hypothesis tested is that the 48 hour rate of major adverse events, Major AE, does not equal 0.40:

 $H_0$ : Major AE = 0.40

vs  $H_a$ : Major  $AE \neq 0.40$ .

under an observed Major AE of 15% at alpha = 0.05.

The power for a one-group, two-sided test for a single proportion was calculated for the test using SAS v 9.4 (SAS Institute, Cary, NC). The SAS code and output are provided in Section 17.

Table 2. Safety Sample Size Parameters

| Alpha | 0.05 |
|-------------------------|-------|
| Sides | 2 |
| Estimated proportion | 0.15 |
| Null proportion $(p_0)$ | 0.40 |
| N | 100 |
| Power | >.999 |

# 2.3 Justification of Effectiveness and Safety Thresholds

**Effectiveness:** A prior study of fibrinolysis identified greater than 0.20 as an appropriate decrease in the RV/LV ratio (Piazza 2015, Fasullo 2011). In this trial a lower limit of 0.2 mean decrease in RV/LV diameter ratio represents a reasonable improvement in effectiveness for this patient population.

**Safety:** Patients with acute pulmonary embolism (PE) have limited alternatives for treatment. While most patients continue to be treated conservatively with anticoagulation alone, high fatality and bleeding rates have been noted. For submassive PE patients, the mortality rate for patients treated with anticoagulation alone was as high as 25% (Konstantinides 2002) and the risk of the major bleeding was less than 8% (Konstantinides 1997). When indicated, more intensive treatment escalation may be required. These include systemic fibrinolysis, emergent surgical embolectomy, and catheter-directed interventions with aspiration or mechanical embolectomy devices.

- Systemic Fibrinolysis is offered to patients who are refractory to anticoagulant therapy. However, systemic thrombolysis is associated with a 20% risk for major bleeding, including a 2 5% risk of hemorrhagic stroke and a mortality rate as high as 11% (Kuo 2015). The clinical deterioration rate for submassive patients treated with systemic fibrinolysis could be as high as 38% (Mehta 2003).
- Emergency Surgical Embolectomy with cardiopulmonary bypass has re-emerged as
  an effective strategy for managing patients with submassive PE with RV dysfunction who
  are not eligible for or are refractory to current standard of care. The mortality rate
  associated with the surgery is as high as 19% (Stein 2012) and in a case series, 3.6% of
  patients had a major bleeding event (Neely 2015).
- Catheter-Directed Intervention is a relatively new treatment option that includes
  catheter-directed fibrinolysis, aspiration or mechanical embolectomy. Early results
  showed this mode of therapy may have promise. According to the limited data available,
  the mortality rate was ~3% (Kuo 2015). The data available on clinical deterioration gives
  a rate of ~3% and ~7% for major bleeding.

In summary, patients with PE who are eligible for the EXTRACT PE trial have few treatment alternatives. These patients are at high risk of morbidity and mortality including those who failed current standard of care. A procedure that is highly effective and has a peri-procedural complications rate of Major Adverse Events with an upper limit of 40% represents a reasonable advance for this patient population. The limited reasonable alternatives justify the proposed safety study success parameter.

This upper limit of 40% was determined from the upper bound of the 95% confidence interval for an estimated major adverse event rate calculated from weighting the published data based on clinical assessment of the importance to the current study.

# 3 Interim Analysis

No interim analyses are planned for the purpose of stopping the study early for success or futility.

An interim sample size review to re-assess the size of the estimated mean and standard deviations of the primary effectiveness variables and the rate of the primary effectiveness safety variables will be performed after  $n_1$  = 50 evaluable patients (i.e. treated only using the Indigo Aspiration System) have primary endpoint data. The sample size will be adjusted accordingly (see section 3.1).

### 3.1 Re-estimation of Sample Size

The initial sample size estimation provides statistical power to demonstrate effectiveness and safety among patients treated only using the Indigo Aspiration System. A potential sample size adjustment is to assure that this trial will have the intended precision. The decision of sample size adjustment will be made based on the estimates of 48 hour mean change in the RV/LV ratio from baseline and 48 hour rate of major adverse events that are calculated for the first 50 evaluable (i.e. treated only using the Indigo Aspiration System) patients with primary endpoint data. The Core Laboratory data and the CEC adjudicated data supersede the investigator-reported data in this sample size re-estimation. Sample size will not be decreased regardless of the results of this evaluation. To warrant the originally intended >80% power of the study at the 0.05 level (2-sided), the evaluable sample size may be increased to a maximum of 300 enrolled patients in order to provide 200 evaluable patients, given expected attrition including use of adjunctive treatments for the purpose of reducing clot burden in pulmonary artery or any use of thrombolytics. The sample size re-estimation will be evaluated for the efficacy endpoint based on the observed interim mean and standard deviation and for the safety endpoint based on the observed interim proportion.

The sample size re-estimation method is based on evaluation of conditional power in relationship to pre-specified decision rules defined by ranges of attainable conditional power values. Only an increase in sample size is possible under this approach when observed conditional power falls within the 'promising zone' as described below (Bhatt 2016, Chen 2004, Cui 1999, Mehta and Pocock 2011, Orloff 2009, PASS 2017).

The conditional power at the interim analysis  $(CP_{\widehat{\delta}_1}(z_1, \widetilde{n_2}))$  can be defined by the following equation from Mehta and Pocock (2011) and PASS (2017):

$$\mathit{CP}_{\widehat{\delta}_1}(z_1,\widetilde{n_2}) = 1 - \Phi\left(\frac{z_{\alpha/2}\sqrt{n_2} - z_1\sqrt{n_1}}{\sqrt{\widetilde{n_2}}} - \frac{z_1\sqrt{\widetilde{n_2}}}{\sqrt{n_1}}\right) + \Phi\left(\frac{-z_{\alpha/2}\sqrt{n_2} - z_1\sqrt{n_1}}{\sqrt{\widetilde{n_2}}} - \frac{z_1\sqrt{\widetilde{n_2}}}{\sqrt{n_1}}\right)$$

where  $\widetilde{n_2}=n_2-n_1$ ,  $z_{\alpha/2}=\Phi^{\text{-1}}(1-\alpha/2)$ , and  $z_1$  is the value of the cumulative Wald statistic as computed at the interim analysis of  $n_1$ = 50 evaluable patients. Define the estimated treatment difference,  $\hat{\delta}_1=\hat{\mu}_1-\mu_0$  or  $\hat{p}_1-p_0$  at interim analysis, where  $\hat{\mu}_1$  and  $\hat{p}_1$  are mean and proportion at interim analysis and  $\mu_0$  and  $p_0$  are the null hypothesis correspondingly.

Our targeted conditional power at the first interim review is 80%, however we pre-specify a range of conditional power values below 80% that would deem our interim results promising and warrant a sample size re-estimation.

Table 3 provides cut-off values from Mehta and Pocock (2011) for the lower bound of the promising zone,  $CP_{min}$ , under some typical two-stage adaptive designs.  $CP_{min}$  is 0.36 (36%) for the parameter choices in this study (Table 5).

Table 3.  $CP_{min}$  cut-off values for some typical two-stage adaptive designs with no early stopping either for efficacy or futility

| Sample siz | e ratios | CP <sub>min</sub> values for targeted | |
|---|---|---|---|
| Sample size ratios | | conditional power | |
| Maximum allowed | At interim look | 80 per cent | 00 per cent |
| $(n_{max}/n_2)$ | $(n_1/n_2)$ | oo per cent | 30 per cent |
| 1.5 | 0.25 | 0.42 | 0.42 |
| 1.5 | 0.5 | 0.41 | 0.41 |
| 1.5 | 0.75 | 0.38 | 0.38 |
| 2 | 0.25 | 0.37 | 0.37 |
| 2 | 0.5 | 0.36 | 0.36 |
| 2 | 0.75 | 0.33 | 0.33 |
| 3 | 0.25 | 0.32 | 0.32 |
| 3 | 0.5 | 0.31 | 0.31 |
| 3 | 0.75 | 0.30 | 0.27 |
| $\infty$ | 0.25 | 0.32 | 0.28 |
| $\infty$ | 0.5 | 0.31 | 0.27 |
| ∞ | 0.75 | 0.30 | 0.25 |

Table 4 summarizes the sample size re-estimation decision based on the conditional power observed at interim analysis. The sample size is re-estimated when the interim conditional power falls within the promising zone of 0.36 to 0.80 (36% to 80%).

Table 4. Sample Size Re-Estimation Decision

| Conditional Power | Decision |
|-------------------|-----------------------------------------------|
| Less than 36% | "Unfavorable Zone" - No change to sample size |
| 36% to 80% | "Promising Zone" - Increase sample size |
| At least 80% | "Favorable Zone" - No change to sample size |

Table 5 provides the parameters used for the sample size re-estimation. We expect that enrollment of up to 300 enrolled patients will provide  $n_{max}$  = 200 evaluable patients. The number of evaluable patients and associated attrition rate including use of adjunctive treatments for the purpose of reducing clot burden in pulmonary artery or any use of thrombolytics will be monitored during the course of the trial until  $n_{max}$  = 200 evaluable patients are achieved.

Table 5. Sample Size Re-Estimation Parameters

| Design Parameters | Value |
|---|---|
| Interim Sample Size, $n_1$ | 50 |
| Cumulative Final Sample Size, $n_2$ | 100 |
| Re-Estimated Cumulative Final Sample Size, n <sub>2</sub> * | Derived Below |
| Pre-specified Maximum Allowable Sample Size, $n_{max}$ | 200 |
| Sample Size Ratio – Maximum Allowed $(n_{max}/n_2)$ | 200/100 = 2 |
| Sample Size Ratio – At Interim Look $(n_1/n_2)$ | 50/100 = 0.5 |
| Incremental Sample Size, $\widetilde{n_2} = n_2 - n_1$ | 50 |
| Re-Estimated Incremental Sample Size, $\tilde{n_2}'$ | Derived Below |
| Estimated Attrition – Monitored during course of trial and | 33% (including an estimated 20% |
| adjusted as appropriate, including an estimated | adjunctive treatment or |
| proportion of subjects receiving adjunctive treatments for | thrombolytic use) |
| the purpose of reducing clot burden in pulmonary artery | |
| or receiving any thrombolytics | |
| Significance Level (Alpha) | 0.05 |

The re-estimated cumulative final sample size  $(n_2^*)$  is computed using the following equation (equation (9) from Mehta and Pocock (2011)) and will be increased by a factor based on a reassessed attrition rate as per the initial sample size calculation:

$$n_2^* = \min(n_2', n_{max})$$
, where  $\tilde{\mathbf{n}}_2'$  satisfies the condition  $\mathit{CP}_{\widehat{\delta}_1}(z_1, \tilde{\mathbf{n}}_2') = 1 - \beta, \beta = 80\%$ , and  $\mathbf{n}_2'$  is the estimated new sample size computed as  $\mathbf{n}_1 + \tilde{\mathbf{n}}_2'$ .

Based on Mehta and Pocock (2011), this condition is satisfied by the function:

$$\tilde{n}_2' = \left(\left[\frac{n_1}{z_1^2}\right]\left[\frac{z_{\alpha/2}\sqrt{n_2}-z_1\sqrt{n_1}}{\sqrt{n_2-n_1}}+z_\beta\right]^2\right)$$
, where  $z_{\alpha/2} = \Phi^{-1}(1-\alpha/2)$ ,  $z_\beta = \Phi^{-1}(1-\beta)$ , and  $z_1$  is the cumulative Wald statistic as computed at the interim analysis of  $n_1$ = 50 patients.

The re-estimation will be conducted for both the effectiveness and safety endpoints and the highest calculated sample size will be utilized to adjust the study enrollment:

$$Re-Estimated\ Cumulative\ Final\ Sample\ Size = \max\{n_{2,Effectiveness}^*, n_{2,Safety}^*\},$$
 subject to  $n_{max}$  = 200.

The SAS code for the calculation of conditional power and sample size re-estimation is provided in Section 17.3.

# 4 Analysis Populations

#### 4.1 Definitions

All primary and secondary effectiveness endpoints will be performed for both the intent-to-treat (ITT) population and per-protocol (PP) population.

 Target Population: Patients presenting with symptoms of acute PE who meet other study entry criteria are eligible for this trial. Enrolled patients will be treated with aspiration thrombectomy by the Indigo<sup>®</sup> Aspiration System.

- Intent-to-Treat Population: All efficacy and safety outcome measures will be analyzed
  under the intent-to-treat (ITT) principle. Under this principle, the ITT population includes
  all patients who signed the informed consent and are enrolled in the study. The data
  from this population will be analysed even if the patient does not follow the protocol until
  completion.
- Modified Intent-to-Treat Population: In addition to the ITT analysis sample, a modified Intent-to-Treat (mITT) sample is defined as a subset of the ITT sample. This population is the primary population for all efficacy parameters. Patients receiving adjunctive treatments for the purpose of reducing clot burden in the pulmonary artery (intraprocedure and up to 48 hours post procedure) or receiving any thrombolytics during the procedure and up to 48-hours post-procedure will be excluded.
- Per-Protocol Population: In addition to the defined ITT analysis sample, a per-protocol
  (PP) sample is defined as a subset of the ITT sample. The per-protocol sample will
  include all enrolled patients who signed the informed consent and do not have significant
  protocol deviations (e.g. eligibility violation or missing primary endpoint assessment).
- Safety Analysis (As Treated) Population: For the safety analysis, a safety sample that is the same as the ITT sample will be examined in which patients will be analyzed according to the actual treatment received.
- Consented but Device Not Introduced: Patients who are consented and have venous
  puncture for the Indigo procedure, but with no component of the Indigo® Aspiration
  System entering the patient's body will be followed through discharge and their safety
  will be summarized separately in the clinical report.

The following additional population definitions apply to this study:

- **Screened:** All patients considered for participation in the study, regardless of whether they have a signed informed consent available.
- Screen Failure: All patients who were evaluated and do not meet the study entry
  criteria, who meet the entry criteria but decline to participate, or who meet the entry
  criteria but have no component of the Indigo System introduced into their body. Patients
  can be screen failed based on general or imaging criteria. These patients may or may
  not have signed an informed consent.

- Enrolled: All patients who have an informed consent form and HIPAA Authorization signed by the subject or LAR, and in whom the Indigo System has been introduced into their body. Informed consent must be obtained prior to enrollment.
- Evaluable: Enrolled patients without use of adjunctive treatments for the purpose of reducing clot burden in pulmonary artery (intra-procedure and up to 48 hours post procedure) and without use of any thrombolytics during the procedure and up to 48hours post-procedure.
- **Completed:** All patients who were enrolled and completed the study Day 30 follow-up or were known to have died prior to Day 30.
- **Early Termination:** All patients who were enrolled but did not complete the study Day 30 follow-up and were not known to have died.

#### 5 Statistical Methods

Summary tables (descriptive statistics and/or frequency tables) will be provided for all baseline variables, effectiveness variables, and safety variables, as appropriate. Continuous variables will be summarized with descriptive statistics (n, mean, standard deviation, range, and median). Frequency counts and percentage of patients within each category will be provided for categorical data. All 95% confidence intervals will be two-sided and presented using the asymptotic or exact intervals for continuous variables and the Wald or Clopper-Pearson intervals for categorical variables. All p-values presented will be two-sided.

#### 6 Baseline Characteristics

Baseline data including, but not limited to demographics, clinical characteristics, and PE characteristics will be summarized using descriptive statistics and the associated 95% confidence intervals.

# 7 Patient Disposition

The number of patients for each of the following categories will be summarized.

- Screen failure patients
- Consented but device not introduced patients
- Enrolled patients

- Evaluable patients
- Patients completing the study; patients not completing the study
- Patients included in the intent to treat population
- Patients included in the modified intent to treat population
- Patients included in the per protocol population
- Patients included in the safety population

### 8 Effectiveness Analysis

## 8.1 Primary Effectiveness Analysis

The primary effectiveness variable is the change in RV/LV ratio at 48 hours. The primary efficacy analysis will be the difference between the baseline and the 48 hours RV/LV diameter ratio. The two-sided 95% confidence interval for the mean difference will be calculated. The primary effectiveness endpoint is met if the lower bound of the confidence interval is >0.2. The confidence interval will be used for testing the primary efficacy hypothesis that the mean change in RV/LV ratio from baseline to 48 hours, RV/LV<sub>change</sub>, does not equal 0.2 at two-sided alpha = 0.05:

 $H_0$ : RV/LV<sub>change</sub> = 0.2

vs  $H_a$ : RV/LV<sub>change</sub>  $\neq$  0.2.

Special consideration will be given to subjects initiating adjunctive treatments for the purpose of reducing clot burden in pulmonary artery (intra-procedure and up to 48 hours post procedure) or receiving any thrombolytics during the procedure and up to 48-hours post-procedure. Such treatments may mask study treatment effect and hence the outcome for these subjects will be conservatively considered an efficacy endpoint failure.

For the purpose of conducting primary effectiveness analyses in our study, the mITT subject data as observed (completer) will be used.

Sensitivity analyses of the primary efficacy endpoint will be performed. Subjects initiating adjunctive treatments for the purpose of reducing clot burden in pulmonary artery (intraprocedure and up to 48 hours post procedure) or receiving any thrombolytics during the procedure and up to 48-hours post-procedure will be analysed as follows for the primary efficacy analyses:

- The change in their RV/LV ratio at 48 hours will be imputed by the worst observed change in RV/LV ratio from the patient population with primary endpoint data
- The change in their RV/LV ratio at 48 hours will be imputed by the best observed change in RV/LV ratio from the patient population with primary endpoint data
- Their observed RV/LV results will be analyzed

For patients who are refractory to other PE treatments pre-procedure, such as EKOS, the change in RV/LV ratio from baseline to 48 hours will not be altered.

The Core Laboratory data supersede the investigator-reported data in all analyses of RV/LV diameter and will be applied to any interim and final primary effectiveness analyses. The primary effectiveness analysis will be performed in the ITT subject population. The analysis based on the Per Protocol (PP) population will be considered as supportive.

# 8.2 Handling of Multiplicity

There will be no adjustment on the primary effectiveness variable since the primary comparison is specified in the protocol. The six subgroup analyses will be considered secondary analyses and will be adjusted using the Bonferroni correction. In the event that the primary endpoint is not met, these subgroup analyses will only be considered as hypothesis generating for future studies.

# 9 Subgroup Analysis

To evaluate the impact of baseline conditions on treatment effect, subgroup analyses will be performed for the primary effectiveness variable, change in the RV/LV ratio, and the primary and secondary safety variables. The subgroups below will be used for these analyses:

- Age
- Gender
- Race/Ethnicity
- Use of IV or IA thrombolytics (tPA) for the purpose of reducing clot burden (intraprocedure and up to 48 hours post procedure)
- Use of IV or IA thrombolytics (tPA) at any time during study follow-up
- Clinical study center
- Operator (e.g. Physician A, Physician B, initial patients treated, subsequent patients treated)

Descriptive statistics will be presented for each subgroup. The subgroup analysis will be conducted using Fisher's exact test, Chi-square test, Wilcoxon rank sum, t-test, Kruskal-Wallis test or ANOVA for univariate analyses and logistic or linear regression for multivariate analyses. These analyses will be performed on the Per Protocol population. The Bonferroni p-value adjustment will be utilized for comparisons between subgroups.

### 10 Safety Analysis

### 10.1 Primary Safety Analysis

The primary safety endpoint is 48 hour major adverse events (device-related death, major bleeding, and peri-procedure device-related SAEs of clinical deterioration, pulmonary vascular injury, and cardiac injury). The proportion of patients who meet the safety endpoint based on this criterion will be calculated and analyzed as a binary variable with each subject counted only once. The two-sided 95% normal distribution confidence interval will be provided for the primary safety endpoint. The CEC data supersede the investigator-reported data in all analyses of adverse events and will be applied to any interim and final safety analyses. The CEC will have final adjudication to determine whether each adverse event satisfies the definition of the primary safety endpoint for the primary safety analysis.

The primary safety endpoint is met if the upper bound of the confidence interval is <40%. The confidence interval will be used for testing the primary safety hypothesis that the rate of 48 hour major adverse events, Major AE, does not equal 40% at two-sided alpha = 0.05:

 $H_0$ : Major AE = 40%

vs  $H_a$ : Major  $AE \neq 40\%$ .

Sensitivity analyses of the primary safety endpoint will be performed for subjects with missing primary endpoint data as described in Section 12.

# 10.2 Secondary Safety Analysis

The secondary safety variables are rates of AEs at 48 hours (device-related death, major bleeding, clinical deterioration, pulmonary vascular injury, and cardiac injury) and AEs at 30 days (any-cause mortality, device-related SAEs, symptomatic PE recurrence). Recurrent PE is defined as symptomatic PE objectively confirmed on contrast-enhanced chest CT, ventilation-perfusion lung scan, or invasive contrast pulmonary angiography. The proportion of patients

who experience a safety event based on these criteria will be calculated along with the associated two-sided 95% confidence interval.

### 10.3 Analysis of Adverse Events

Tabulations of adverse events will be presented with descriptive statistics at baseline hospitalization and follow-up visits. Adverse event incidence rates will be summarized by category and seriousness of the adverse event. Each subject will be counted only once within a category by using the adverse event with the highest seriousness within each category.

All information pertaining to adverse events noted during the study will be listed by subject, detailing verbatim given by the investigator, category, date of onset, date of resolution, causality and severity. The onset of adverse events will also be shown relative (in number of days) to the day of procedure.

A tabulation of Serious Adverse Events (SAEs) will be provided by subject.

The specific categories analyzed will be those that are reported by at least three (3) percent of the patients. The CEC adjudicated data supersedes the investigator reported data in all analyses of adverse events.

# **10.4 Handling of Multiplicity**

There will be no adjustment for multiple comparisons on the primary safety variable since the primary comparison is specified in the protocol. The subgroup safety analyses will be considered secondary and will be adjusted using the Bonferroni correction.

# 10.5 Analysis of Deaths

The Kaplan-Meier product-limit method will be the primary method utilized to assess the mortality rate. With the date of procedure set at Day 0, any death occurring on or before calendar day 30 will be counted as a death. If clinical assessment is missing for a patient who has not died, the patient will be censored at the last follow-up date. Patients who are alive at day 30 will be censored at day 30. The time to death will be plotted with confidence intervals at monthly intervals.

Additionally, the death data will be presented as 30 Day binary deaths. The number of deaths will be presented with the 95% confidence interval.

### 11 Pooling Across Centers

The clinical study will be conducted under a common protocol for each investigational center with the intention of pooling the data for analysis. Every effort will be made to promote consistency in study execution at each investigational center. Analyses will be presented using data pooled across centers. Appropriate stratification and multivariate techniques, including random effects, contingency tables and logistic regression for binary outcomes, analysis of variance for continuous measures, and proportional hazards regression for time-to-event outcomes, will be used to assess differences between study centers to justify pooling data across centers. Centers with fewer than 10 patients may be combined and treated as one site in the pooling analysis, up to a limit of 30 patients per pooled site.

# 12 Lost to Follow-Up and Missing Data

For sensitivity purposes, the following additional analyses will be conducted for the primary efficacy endpoint:

- For those patients without any observations after procedure:
  - Their 48-hour post-procedure observations will be imputed by baseline scores and included in an analysis.
  - The change in their RV/LV ratio at 48 hours will be imputed using the worst observed change in RV/LV ratio from the patient population with primary endpoint data.
  - The change in their RV/LV ratio at 48 hours will be imputed using the best observed change in RV/LV ratio from the patient population with primary endpoint data.

Sensitivity analyses of the primary safety endpoint will be performed for subjects with missing primary safety endpoint at 48 hour follow-up as follows:

- The subjects will be excluded from analysis
- Their primary safety outcome will be imputed using the worst clinical scenario assuming the subject experienced a primary safety event
- Their primary safety outcome will be imputed using the best clinical scenario assuming the subject did not experience a primary safety event

 If needed, a tipping point analysis will be conducted in which the missing data will be replaced with values such that the upper bound of the confidence interval is greater than 40%

### 13 Blinding

The Penumbra Inc. clinical team responsible for the conduct of the study, the investigator, study center personnel, core laboratory and clinical events committee will not be blinded to each patient's treatment throughout the course of the study.

#### 14 Committees

#### 14.1 Clinical Events Committee (CEC)

A CEC will adjudicate adverse events for causality and attribution.

### 14.2 Data Safety Monitoring Board (DSMB)

The DSMB will review the overall safety of the trial.

#### 14.3 Core Lab

An independent Core Lab will review and score imaging scans for RV/LV ratio.

# 15 Changes to Planned Analyses

All changes to the statistical analysis plan (SAP) will be documented in a revised SAP or the clinical study report.

### 16 References

Agresti, A. (2012). Categorical Data Analysis (Third Edition). John Wiley & Sons.

Aklog, L., Williams, C. S., Byrne, J. G., & Goldhaber, S. Z. (2002). Acute pulmonary embolectomy. *Circulation*, *105*(12), 1416-1419.

Bajaj, N. S., Kalra, R., Arora, P., Ather, S., Guichard, J. L., Lancaster, W. J., ... & Clark, D. T. (2016). Catheter-directed treatment for acute pulmonary embolism: Systematic review and single-arm meta-analyses. *International Journal of Cardiology*, *225*, 128-139.

Becattini, C., Agnelli, G., Salvi, A., Grifoni, S., Pancaldi, L. G., Enea, I., ... & TIPES Study Group. (2010). Bolus tenecteplase for right ventricle dysfunction in hemodynamically stable patients with pulmonary embolism. *Thrombosis research*, *125*(3), e82-e86.

Bhatt, D. L., & Mehta, C. (2016). Adaptive designs for clinical trials. *New England Journal of Medicine*, *375*(1), 65-74.

Chen, Y. H., DeMets, D. L., & Gordon Lan, K. K. (2004). Increasing the sample size when the unblinded interim result is promising. Statistics in medicine, 23(7), 1023-1038.

Cui, L., Hung, H. M., & Wang, S. J. (1999). Modification of sample size in group sequential clinical trials. Biometrics, 55(3), 853-857.

Chow, S.C., Shao, J., Wang, H. (2008). <u>Sample Size Calculations in Clinical Research (Second Edition</u>). Boca Raton, Chapman & Hall/CRC.

Fasullo, S., Scalzo, S., Maringhini, G., Ganci, F., Cannizzaro, S., Terrazzino, G., ... & Cangemi, D. (2011). Six-month echocardiographic study in patients with submassive pulmonary embolism and right ventricle dysfunction: comparison of thrombolysis with heparin. *The American journal of the medical sciences*, *341*(1), 33-39.

Gallotta, G., Palmieri, V., Piedimonte, V., Rendina, D., De Bonis, S., Russo, V., ... & Di Minno, G. (2008). Increased troponin I predicts in-hospital occurrence of hemodynamic instability in patients with sub-massive or non-massive pulmonary embolism independent to clinical, echocardiographic and laboratory information. *International journal of cardiology*, *124*(3), 351-357.

Garcia, M. J., Lookstein, R., Malhotra, R., Amin, A., Blitz, L. R., Leung, D. A., ... & Soukas, P. A. (2015). Endovascular management of deep vein thrombosis with rheolytic thrombectomy: final report of the prospective multicenter PEARL (Peripheral Use of AngioJet Rheolytic Thrombectomy with a Variety of Catheter Lengths) registry. *Journal of Vascular and Interventional Radiology*, 26(6), 777-785.

Greelish, J. P., Leacche, M., Solenkova, N. S., Ahmad, R. M., & Byrne, J. G. (2011). Improved midterm outcomes for type A (central) pulmonary emboli treated surgically. *The Journal of thoracic and cardiovascular surgery*, *142*(6), 1423-1429.

Hollander, M., Wolfe, D. A., & Chicken, E. (2013). <u>Nonparametric Statistical Methods (Second Edition)</u>. John Wiley & Sons.

Kalbfleisch, J. D., & Prentice, R. L. (2011). <u>The Statistical Analysis of Failure Time Data</u> (Second Edition). John Wiley & Sons.

Kline, J. A., Nordenholz, K. E., Courtney, D. M., Kabrhel, C., Jones, A. E., Rondina, M. T., ... & Hernandez, J. (2014). Treatment of submassive pulmonary embolism with tenecteplase or placebo: cardiopulmonary outcomes at 3 months: multicenter double-blind, placebo-controlled randomized trial. *Journal of Thrombosis and Haemostasis*, *12*(4), 459-468.

Konstantinides, S., Geibel, A., Olschewski, M., Heinrich, F., Grosser, K., Rauber, K., ... & Kasper, W. (1997). Association between thrombolytic treatment and the prognosis of hemodynamically stable patients with major pulmonary embolism. *Circulation*, *96*(3), 882-888.

Konstantinides, S., Geibel, A., Heusel, G., Heinrich, F., & Kasper, W. (2002). Heparin plus alteplase compared with heparin alone in patients with submassive pulmonary embolism. *New England Journal of Medicine*, *347*(15), 1143-1150.

Kucher, N., Printzen, G., & Goldhaber, S. Z. (2003). Prognostic role of brain natriuretic peptide in acute pulmonary embolism. *Circulation*, *107*(20), 2545-2547.

Kucher, N., Boekstegers, P., Müller, O., Kupatt, C., Beyer-Westendorf, J., Heitzer, T., ... & Greif, M. (2014). Randomized controlled trial of ultrasound-assisted catheter-directed thrombolysis for acute intermediate-risk pulmonary embolism. *Circulation*, CIRCULATIONAHA-113.

Kuo, W. T., Banerjee, A., Kim, P. S., DeMarco, F. J., Levy, J. R., Facchini, F. R., ... & Rosenberg, J. K. (2015). Pulmonary embolism response to fragmentation, embolectomy, and catheter thrombolysis (PERFECT): initial results from a prospective multicenter registry. *CHEST Journal*, *148*(3), 667-673.

Leacche, M., Unic, D., Goldhaber, S. Z., Rawn, J. D., Aranki, S. F., Couper, G. S., ... & Byrne, J. G. (2005). Modern surgical treatment of massive pulmonary embolism: results in 47 consecutive patients after rapid diagnosis and aggressive surgical approach. *The Journal of Thoracic and Cardiovascular Surgery*, 129(5), 1018-1023.

Mehta, C. R., & Pocock, S. J. (2011). Adaptive increase in sample size when interim results are promising: a practical guide with examples. *Statistics in medicine*, *30*(28), 3267-3284.

Mehta, N. J., Jani, K., & Khan, I. A. (2003). Clinical usefulness and prognostic value of elevated cardiac troponin I levels in acute pulmonary embolism. *American heart journal*, *145*(5), 821-825.

Meyer, G., Vicaut, E., Danays, T., Agnelli, G., Becattini, C., Beyer-Westendorf, J., ... & Dellas, C. (2014). Fibrinolysis for patients with intermediate-risk pulmonary embolism. *New England Journal of Medicine*, *370*(15), 1402-1411.

Neely, R. C., Byrne, J. G., Gosev, I., Cohn, L. H., Javed, Q., Rawn, J. D., ... & Leacche, M. (2015). Surgical embolectomy for acute massive and submassive pulmonary embolism in a series of 115 patients. *The Annals of thoracic surgery*, *100*(4), 1245-1252.

Orloff, J., Douglas, F., Pinheiro, J., Levinson, S., Branson, M., Chaturvedi, P., ... & Patel, N. (2009). The future of drug development: advancing clinical trial design. *Nature reviews. Drug discovery*, *8*(12), 949.

PASS sample size software. Conditional Power of One-Sample T-Tests. Retrieved from <a href="https://ncss-wpengine.netdna-ssl.com/wp-content/themes/ncss/pdf/">https://ncss-wpengine.netdna-ssl.com/wp-content/themes/ncss/pdf/</a> Procedures/PASS/Conditional Power of One-Sample T-Tests.pdf.

PASS sample size software. Conditional Power of One Proportion Tests. Retrieved from <a href="https://ncss-wpengine.netdna-ssl.com/wp-content/themes/ncss/pdf/Procedures/PASS/">https://ncss-wpengine.netdna-ssl.com/wp-content/themes/ncss/pdf/Procedures/PASS/</a> Conditional Power of One Proportion Tests.pdf.

Piazza, G., Hohlfelder, B., Jaff, M. R., Ouriel, K., Engelhardt, T. C., Sterling, K. M., ... & Goswami, N. (2015). A prospective, single-arm, multicenter trial of ultrasound-facilitated, catheter-directed, low-dose fibrinolysis for acute massive and submassive pulmonary embolism: The SEATTLE II Study. *JACC: Cardiovascular Interventions*, *8*(10), 1382-1392.

Pieralli, F., Olivotto, I., Vanni, S., Conti, A., Camaiti, A., Targioni, G., ... & Berni, G. (2006). Usefulness of bedside testing for brain natriuretic peptide to identify right ventricular dysfunction and outcome in normotensive patients with acute pulmonary embolism. *The American journal of cardiology*, *97*(9), 1386-1390.

Quiroz, R., Kucher, N., Schoepf, U. J., Kipfmueller, F., Solomon, S. D., Costello, P., & Goldhaber, S. Z. (2004). Right ventricular enlargement on chest computed tomography. *Circulation*, *109*(20), 2401-2404.

Stein, P. D., & Matta, F. (2012). Case fatality rate with pulmonary embolectomy for acute pulmonary embolism. *The American journal of medicine*, *125*(5), 471-477.

Stokes, M. E., Davis, C. S., & Koch, G. G. (2012). <u>Categorical Data Analysis Using SAS® (Third Edition)</u>. Cary, NC, SAS Institute

### 17 SAS Code

# **17.1 Primary Efficacy Power Calculation**

#### 17.1.1 Code

title1 "Efficacy Power Calculation with mean of 0.42 and SD of 0.36";

proc power;
onesamplemeans
nullmean = 0.2
mean = .42
stddev = 0.36
power=.
ntotal = 100;
run;

#### 17.1.2 Output

| The POWER Procedure |
|-----------------------------|
| THE FOWLKT TOCCULE |
| One-Sample t Test for Mean |
| One-sample t lest for weari |

| Fixed Scenario Elements | |
|-------------------------|--------|
| Distribution | Normal |
| Method | Exact |
| Null Mean | 0.2 |
| Mean | 0.42 |
| Standard Deviation | 0.36 |
| Total Sample Size | 100 |
| Number of Sides | 2 |
| Alpha | 0.05 |

Computed Power Power >.999

## **17.2 Primary Safety Power Calculation**

#### 17.2.1 Code

title1 "Safety Power Calculation with a safety proportion of 0.15 and a null proportion of 0.40"; proc power;
onesamplefreq test = Z method = normal
nullproportion = 0.40
proportion = 0.15
ntotal = 100
power = .;
run;

#### 17.2.2 Output

# The POWER Procedure Z Test for Binomial Proportion

| Fixed Scenario Elements | |
|----------------------------|----------------------|
| Method | Normal approximation |
| Null Proportion | 0.4 |
| <b>Binomial Proportion</b> | 0.15 |
| Total Sample Size | 100 |
| Variance Estimate | Null Variance |
| Number of Sides | 2 |
| Alpha | 0.05 |



### 17.3 Sample Size Re-Estimation Calculation

```
macro for sample size re-estimation based on promising zone: for one sample mean variables;
mu0 = null mean
mu1 hat = observed interim mean
sigma1 hat = observed interim standard deviation
cp min = minimum conditional power for promising zone
power = targeted conditional power
n1 = interim sample size
n2 = cumulative final sample size
nmax = pre-specified maximum allowable sample size
drop = estimated attrition
cp = conditional power
size = re-estimated cumulative final sample size
enroll = total enrollment including dropouts
test = z test value based on new sample size (if required to be increased)
new alpha = p-value checked based on new n
***/
%macro simulation(mu0=,cp_min=,power=,n1=,n2=,nmax=,drop=);
 data a:
  length zone $30 estimate $50;
  alpha = 0.05;
  n2 tilde = &n2 - &n1;
        do mu1 hat = 0.225 to 0.8 by 0.01;
        do sigma1_hat = 0.3 to 0.95 by 0.01;
        za = quantile('NORMAL',1-alpha/2);
   zb = quantile('NORMAL',&power);
   se_delta1_hat = sigma1_hat / sqrt(&n1);
   delta1 hat = mu1 hat - &mu0;
   z1 = delta1 hat / se delta1 hat;
   cp u = 1 - cdf('NORMAL', (za * sqrt(&n2) - z1 * sqrt(&n1)) / sqrt(n2 tilde) - (z1 * sqrt(n2 tilde)) /
        cp I = cdf('NORMAL', (-za * sqrt(&n2) - z1 * sqrt(&n1)) / sqrt(n2 tilde) - (z1 * sqrt(n2 tilde)) /
sqrt(&n1));
        cp = cp u + cp I;
        /*** conditions to check if value falls within promising zone ***/
        if cp ge &cp min and cp le &power then do;
         zone = "Promising Zone";
         estimate = "Sample size should be increased";
         n2 tilde prime = ceil((&n1 / z1 ** 2) * ((za * sqrt(&n2) - z1 * sqrt(&n1)) / sqrt(&n2 - &n1) + zb) **
2);
   n2 prime = &n1 + n2 tilde prime;
   size = min(n2 prime, &nmax);
   enroll = ceil(size/(1-&drop));
         test = delta1 hat/(sigma1 hat/sqrt(size));
   power1 = cdf('NORMAL',test-za) + cdf('NORMAL',-test-za);
   new_alpha = 2 * (1 - cdf('NORMAL', abs(test)));
        end;
         if cp gt &power then do;
         zone = "Favorable zone";
```

```
estimate = "Sample size should not be increased";
        size = &n2:
        enroll = ceil(size/(1-&drop));
        test = delta1 hat/(sigma1 hat/sqrt(&n2));
        power1 = cdf('NORMAL'.test-za) + cdf('NORMAL'.-test-za):
        new_alpha = 2 * (1 - cdf('NORMAL', abs(test)));
        end;
        if cp lt &cp min then do;
        zone = "Unfavorable zone";
        estimate = "Sample size should not be increased";
        size= &n2:
        enroll = ceil(size/(1-&drop));
        test = delta1 hat/(sigma1 hat/sqrt(&n2));
   power1 = cdf('NORMAL',test-za) + cdf('NORMAL',-test-za);
        new_alpha = 2 * (1 - cdf('NORMAL', abs(test)));
   end:
        output;
       end;
 end;
 keep mu1_hat sigma1_hat za alpha size enroll zone estimate power1 new_alpha cp;
label
       mu1 hat = "Observed Interim Mean"
       sigma1 hat = "Observed Interim SD"
       za = "Za"
       alpha = "Alpha"
       size = "Re-Estimated Cumulative Final Sample Size"
       enroll = "Re-Estimated Cumulative Final Enrolled Sample Size (To Accommodate Dropout)"
       zone = "Zone"
       estimate = "Decision"
       power1 = "Power"
       new alpha = "Interim P-Value with this Scenario"
       cp = "Conditional Power";
 run;
%mend:
%simulation(mu0=0.2,cp min=0.36,power=0.8,n1=50,n2=100,nmax=200,drop=0.33);
macro for sample size re-estimation based on promising zone: for one sample proportion variables;
p0 = null proportion
p1 hat = observed interim proportion
sigma1 hat = observed interim standard deviation
cp min = minimum conditional power for promising zone
power = targeted conditional power
n1 = interim sample size
n2 = cumulative final sample size
nmax = pre-specified maximum allowable sample size
drop = estimated attrition
cp = conditional power
size = re-estimated cumulative final sample size
enroll = total enrollment including dropouts
test = z test value based on new sample size (if required to be increased)
new alpha = p-value checked based on new n
```

```
%macro psimulation(p0=,cp_min=,power=,n1=,n2=,nmax=,drop=);
 data a prop:
  length zone $30 estimate $50;
  alpha = 0.05;
  n2 tilde = &n2 - &n1;
        do p1_hat = 0.1 \text{ to } 0.7 \text{ by } 0.025;
         sigma1 hat = sqrt(p1 hat*(1-p1 hat));
   za = quantile('NORMAL',1-alpha/2);
   zb = quantile('NORMAL',&power);
   se delta1 hat = sigma1 hat / sgrt(&n1);
   delta1 hat = p1 hat - &p0;
   z1 = delta1 hat / se delta1 hat;
   cp u = 1 - cdf('NORMAL', (za * sqrt(&n2) - z1 * sqrt(&n1)) / sqrt(n2 tilde) - (z1 * sqrt(n2 tilde)) /
sqrt(&n1));
         cp_I = cdf('NORMAL', (-za * sqrt(&n2) - z1 * sqrt(&n1)) / sqrt(n2_tilde) - (z1 * sqrt(n2_tilde)) /
sqrt(&n1));
        cp = cp_u + cp_l;
         /*** conditions to check if value falls within promising zone ***/
         if cp ge &cp min and cp le &power then do;
         zone = "Promising Zone";
         estimate = "Sample size should be increased";
         n2 tilde prime = ceil((&n1 / z1 ** 2) * ((za * sqrt(&n2) - z1 * sqrt(&n1)) / sqrt(&n2 - &n1) + zb) **
2);
   n2 prime = &n1 + n2 tilde prime;
   size = min(n2 prime, &nmax);
   enroll = ceil(size/(1-&drop));
   test = delta1_hat/(sigma1_hat/sqrt(size));
         power1 = cdf('NORMAL',test-za) + cdf('NORMAL',-test-za);
         new alpha = 2 * (1 - cdf('NORMAL', abs(test)));
         end:
         else if cp gt &power then do;
         zone = "Favorable zone":
         estimate = "Sample size should not be increased";
         size =&n2:
         enroll = ceil(size/(1-&drop));
         test = delta1 hat/(sigma1 hat/sqrt(&n2));
         power1 = cdf('NORMAL',test-za) + cdf('NORMAL',-test-za);
         new_alpha = 2 * (1 - cdf('NORMAL', abs(test)));
         end;
         else if cp It &cp min then do;
         zone = "Unfavorable zone";
         estimate = "Sample size should not be increased";
         size= &n2:
         enroll = ceil(size/(1-&drop));
         test = delta1 hat/(sigma1 hat/sqrt(&n2));
         power1 = cdf('NORMAL',test-za) + cdf('NORMAL',-test-za);
   new_alpha = 2 * (1 - cdf('NORMAL', abs(test)));
        end:
                 output;
   end;
          keep p1 hat sigma1 hat za alpha size enroll zone estimate power1 new alpha cp;
```

```
label

p1_hat = "Observed Interim Proportion"
sigma1_hat = "Observed Interim SD"
Za = "Za"
alpha = "Alpha"
size = "Re-Estimated Cumulative Final Sample Size"
enroll = "Re-Estimated Cumulative Final Enrolled Sample Size (To Accommodate Dropout)"
zone = "Zone"
estimate = "Decision"
power1 = "Power"
new_alpha = "Interim P-value with this Scenario"
cp = "Conditional Power";
run;
%mend;
%psimulation(p0=0.4,cp_min=0.36,power=0.8,n1=50,n2=100,nmax=200,drop=0.33)
```